CLINICAL TRIAL: NCT01384643
Title: Effect of Propofol on Renal Injury in Patients Undergoing Valvular Heart Surgery: A Prospective, Randomized Controlled Trial
Brief Title: Effect of Propofol on Renal Injury in Patients Undergoing Valvular Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1-2011-0007
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Heart Valve Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol group (Experimental)
  Interventions: Drug: Propofol
- Control group (Placebo Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Induction of anesthesia: Propofol 1 mg/kg, sufentanil 1.0-3.0 µg/kg and rocuronium 50 mg IV Maintenance of anesthesia (pre CPB): Propofol 120-600 µg ∙ kg-1 ∙ h-1 , sufentanil 0.15-0.3 µg ∙ kg-1 ∙ h-1, vecuronium 8-10 mg/h IV infusion Maintenance of anesthesia (during CPB): Propofol 120-600 µg ∙ kg-1 ∙ h-1 IV infusion Weaning from CPB: Sufentanil 50 µg IV Maintenance of anesthesia (post CPB): Propofol 120-600 µg ∙ kg-1 ∙ h-1 , sufentanil 0.15-0.3 µg ∙ kg-1 ∙ h-1, vecuronium 8-10 mg/h IV infusion Propofol infusion rate is titrated using bispectral index (40-60).

SUMMARY:
Ischemia/reperfusion (I/R)-induced acute kidney injury is a serious complication affecting patient outcome following cardiovascular surgeries. Propofol, an intravenously administered anesthetic with antioxidant properties, protects organs from I/R injury. This study aimed to investigate the ability of propofol to protect kidneys against I/R injury in the patients undergoing valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing valvular heart surgery.
* Age: 20~75.

Exclusion Criteria:

* Emergency operation.
* Patients with vitamin E or vitamin C within 5 days before surgery.
* Patients with preoperative C-reactive protein (CRP) > 16 mg/L.
* Patients with serum creatinine ≥ 2.0 mg/dL
* Patients under hemodialysis.
* Patients with acute myocardial infarction within 1 week before surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Serum creatinine | incidence of AKI during 48 hours after the surgery incidence of AKI
  Comparison of serum creatinine elevation after surgery between Propofol and Control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea